CLINICAL TRIAL: NCT01482013
Title: A Double-blind, Randomized, Placebo-controlled, Phase I , Multiple-dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Orally-administered HPP854 in Subjects With Mild Cognitive Impairment or a Diagnosis of Mild Alzheimer's Disease
Brief Title: Safety Study of HPP854 in Subjects With Mild Cognitive Impairment or a Diagnosis of Mild Alzheimer's Disease
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: High Point Pharmaceuticals, LLC. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HPP854-104
Record Dates: First submitted 2011-11-10; First posted 2011-11-30 (Estimated); Last update posted 2012-08-30 (Estimated); Status verified 2012-08

CONDITIONS: Mild Alzheimer's Disease; Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- HPP854 (Experimental): Oral HPP854 once a day for 28 days.
  Interventions: Drug: HPP854
- Placebo (Placebo Comparator): Oral, placebo once a day for 28 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HPP854 — Oral, once a day for 28 days.
  Arms: HPP854
Drug: Placebo — Oral, once a day for 28 days.
  Arms: Placebo

SUMMARY:
This is a safety and tolerability study investigating the effect of HPP854 in subjects with mild cognitive impairment or a diagnosis of mild Alzheimer's disease. The study will assess the pharmacokinetic and pharmacodynamic relationships of HPP854 in plasma, pharmacodynamic relationship in cerebral spinal fluid and plasma concentration profiles for Amyloid-Beta.

ELIGIBILITY:
Inclusion Criteria:

* Medical history for at least 6 months prior to screening of mild cognitive impairment with a Mini Mental State Exam (MMSE) score between 20 and 26 or diagnosis of mild Alzheimer's disease;
* Must be able to swallow dose of study medication;
* Body Mass Index (BMI) between 18.0 and 35.0; and
* Subject and Project Partner are willing to participate and agree to comply with all study requirements.

Exclusion Criteria:

* Blood pressure > 160 mmHg (systolic) and > 90 mmHg (diastolic);
* Received HPP854 in a previous trial;
* Participation in another clinical trial involving any marketed or investigational drug within 30 days of screening and until after the final study visit.
* Current evidence or history within the last 3 years of a neurological or psychiatric illness that could contribute to dementia including but not limited to: anxiety, epilepsy, focal brain lesion, Parkinson's disease, seizure disorder, or head injury with loss of consciousness and alcohol or substance abuse;
* Clinically significant cardiovascular, cerebrovascular disease, diabetic condition, hematologic, renal hepatic, pulmonary, endocrine, neurological, coagulation disorder;
* History or presence of cancer except for non melanoma skin cancer. Subjects with a history of prostate cancer stable for > 3 yrs with no active treatment for > 3 years prior to Screening may be considered for eligibility;
* Use of the following medications/therapy from 14 days before dosing until after the Final Visit: anti-cholinergic, tricyclic antidepressants, lithium, typical or atypical antipsychotic medications, anticonvulsant medications, immunosuppressive agents, oral corticosteroids, and radiotherapy;
* HbA1C > 6.5 % at the Screening Visit;
* Vitamin B12 level < 211 pg/mL at the Screening Visit;
* Any suicidal risk determined by C-SSRS administered by a study staff member appropriately certified for administration of the scale (Baseline/Screening, Phase 1 Study Version) at Screening Visit, Day -6 or Day -1;
* A score of 15 or more on the modified Geriatric Depression Scale (GDS); and
* A score of 5 or more on the Hashinski Ischemic Scale (Rosen modification.
* Contraindications of MRI including: Metallic fragments, clips or devices in the brain, eye, spinal canal, etc; Cardiac pacemakers, insulin pumps, neurostimulators, cochlear implants, etc.
* Contraindications for blood or CSF sampling, including: Bleeding disorder or taking anticoagulants/antiplatelet, chronic active infection.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2011-10; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Number of Participant Adverse Events | Day 1 to Day 30

SECONDARY OUTCOMES:
Evaluation of participant plasma HPP854 concentrations | Day 1 to Day 30
Change in cerebrospinal fluid concentration of Amyloid-Beta | Day -6 to Day 35

CONTACTS AND LOCATIONS:
Overall Officials: Robert Hernandez, Ph.D., Study Director — High Point Pharmaceuticals, LLC.
Locations (3):
- United States (3):
  - Elite Research Institute, Miami, Florida
  - Duke Clinical Research Unit, Durham, North Carolina
  - High Point Clinical Trials Center, High Point, North Carolina